CLINICAL TRIAL: NCT06942169
Title: The Effects of Mindfulness-Based Self-Compassion Training for Menopausal Women on Their Genital Self-Image and Self-Anger
Brief Title: Mindfulness-Based Self-Compassion Training for Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Aysel AKBENIZ, Assoc. Prof. Dr., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/4613
Record Dates: First submitted 2025-04-08; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Menopausal; Crisis; Self-Compassion; Image, Body; Anger
Keywords: Self-Compassion; anger; Menopause; Image, Body; mindfulness

STUDY DESIGN:
Intervention Model Description: The study was executed in the form of a randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor did not know whose study or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Self-Compassion Training (Experimental): Mindfulness-Based Self-Compassion Training is a very comprehensive approach that addresses the awareness and acceptance of individuals towards their bodies, as well as encouraging them to live a conscious life. Studies found that self-compassion increases well-being during menopause.
  Interventions: Behavioral: Mindfulness-Based Self-Compassion Training
- No intervention (No Intervention): No intervention was applied to menopausal women in the control group.

INTERVENTIONS:
Behavioral: Mindfulness-Based Self-Compassion Training — Mindfulness-Based Self-Compassion Training is a very comprehensive approach that addresses the awareness and acceptance of individuals towards their bodies, as well as encouraging them to live a conscious life. Studies found that self-compassion increases well-being during menopause (Brown, 2015; Arab et al., 2020). Psychiatric nursing is a special field that works to evaluate, diagnose, and enhance mental health in every area where people are present.
  Arms: Mindfulness-Based Self-Compassion Training

SUMMARY:
This study was conducted to determine the effects of mindfulness-based self-compassion training for menopausal women on their genital self-image and self-anger.

Materials and Methods: This study was randomized with 126 menopausal women (study group n=63, control group n=63) between June 2024 and February 2025. Mindfulness-Based Self-Compassion Training (MBSCT) was applied in groups of 10 and 11 participants, twice a week, for 8 sessions of 40 minutes. Data were obtained using the Personal Information Form, Female Genital Self-Image Scale (FGSIS), and DSM-V Level II Anger Scale.

Research Hypotheses:

H1: MBSCT applied to menopausal women enhances the genital self-image of individuals.

H2: MBSCT applied to menopausal women reduces individuals' self-anger.

DETAILED DESCRIPTION:
The menopausal period is a period of physical and mental changes in which the body enters the aging process and the functionality of the genital organs decreases. During this period, women face negative body image, low genital self-image, and inadequate sexual functions. Perceived negative body image can lead to consequences such as low genital self-image and sexual dissatisfaction.

Mindfulness-Based Self-Compassion Training is a very comprehensive approach that addresses the awareness and acceptance of individuals towards their bodies, as well as encouraging them to live a conscious life. Studies found that self-compassion increases well-being during menopause . Psychiatric nursing is a special field that works to evaluate, diagnose, and enhance mental health in every area where people are present. However, midwifery has a wide service area with the priority of preventive health services; primarily women's health, and the duties of evaluating, diagnosing, enhancing, and rehabilitating the physical and psychological health of the whole family. In light of this information, increasing the mindfulness and self-compassion levels of women in menopause may increase the place of women who "age" healthily and therefore mentally healthy elderly women, in society and may make a significant contribution to protecting and improving the mental health of society. Since the literature review revealed a gap in the literature regarding these areas for women in the menopausal period, this study was conducted to determine the effects of mindfulness-based self-compassion training for menopausal women on their genital self-image and self-anger.

ELIGIBILITY:
Inclusion Criteria:

* Being between 45 and 70 years old
* Having no hearing problems
* Being at menopause in the last year
* Having no psychiatric illness
* Having natural menopause
* Not receiving hormone replacement therapy.

Exclusion Criteria:

* Those who did not attend two or more training sessions during the study were excluded from the study.
* Those who entered menopause surgically and received hormone/replacement therapy during the process were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Female Genital Self-Image Scale (FGSIS) | baseline and after 8 weeks
  The Female Genital Self-Image Scale (FGSIS) was developed by Herbenick and Reece (2010) in the United States to measure women's genital self-perceptions.

SECONDARY OUTCOMES:
DSM-V Level 2 Anger Scale | baseline and after 8 weeks
  The Turkish validity and reliability of the Level II Anger Scale prepared by the American Psychiatric Association for DSM-V was conducted by Çöldür et al. (2017). The DSM-V Level II Anger Scale is a five-item self-report scale used to measure the level of self-anger in adults and provides a practical measurement. Each item asks the individual to rate the severity of their anger at themselves over the last 7 days. Scale scoring ranges from 5 to 25.

CONTACTS AND LOCATIONS:
Locations (1):
- Family Health Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
To conduct the study, approval was obtained from the Scientific Research and Publication Ethics Committee of XXX University (APPROV NO: 2023/4613) and legal permission was obtained from the institutions where the study would be conducted. The purpose of the study was explained to the patients included in the study and their questions were answered. It was explained to the patients that the information they provided would be kept confidential, would not be used anywhere else, and that they had the right to withdraw from the study at any time. Before starting the study, the purpose of the study was explained to the patients and their relatives, and their verbal and written permissions were obtained.
Supporting Information: ICF
Time Frame: Before starting the study, the purpose of the study was explained to the patients and their relatives, and their verbal and written permissions were obtained.
Access Criteria: ANYONE PARTICIPATING IN THE RESEARCH WILL BE ABLE TO ACCESS IT.

REFERENCES:
- [Background] Crego A, Yela JR, Riesco-Matias P, Gomez-Martinez MA, Vicente-Arruebarrena A. The Benefits of Self-Compassion in Mental Health Professionals: A Systematic Review of Empirical Research. Psychol Res Behav Manag. 2022 Sep 14;15:2599-2620. doi: 10.2147/PRBM.S359382. eCollection 2022. PMID 36133626
- [Result] Algars M, Huang L, Von Holle AF, Peat CM, Thornton LM, Lichtenstein P, Bulik CM. Binge eating and menstrual dysfunction. J Psychosom Res. 2014 Jan;76(1):19-22. doi: 10.1016/j.jpsychores.2013.11.011. Epub 2013 Nov 28. PMID 24360136
- [Result] de Salis I, Owen-Smith A, Donovan JL, Lawlor DA. Experiencing menopause in the UK: The interrelated narratives of normality, distress, and transformation. J Women Aging. 2018 Nov-Dec;30(6):520-540. doi: 10.1080/08952841.2018.1396783. Epub 2017 Nov 2. PMID 29095126
- [Result] Guest E, Costa B, Williamson H, Meyrick J, Halliwell E, Harcourt D. The effectiveness of interventions aiming to promote positive body image in adults: A systematic review. Body Image. 2019 Sep;30:10-25. doi: 10.1016/j.bodyim.2019.04.002. Epub 2019 May 9. PMID 31077956
- [Result] Handy AB, Greenfield SF, Yonkers KA, Payne LA. Psychiatric Symptoms Across the Menstrual Cycle in Adult Women: A Comprehensive Review. Harv Rev Psychiatry. 2022 Mar-Apr 01;30(2):100-117. doi: 10.1097/HRP.0000000000000329. PMID 35267252
- [Result] Kim MK, Ahn CW, Nam JS, Kang S, Park JS, Kim KR. Association between nonalcoholic fatty liver disease and coronary artery calcification in postmenopausal women. Menopause. 2015 Dec;22(12):1323-7. doi: 10.1097/GME.0000000000000503. PMID 26154274
- Available data/document: Informed Consent Form — https://www.inonu.edu.tr/sagbilgiretik/menu/12561/bilgilendirici-onam-formu — Informed consent is the process by which a patient freely and consciously gives consent after receiving sufficient information about the medical procedure, treatment or intervention to be applied to him/her. The written form of this process is the Informed Consent Form.